CLINICAL TRIAL: NCT02643927
Title: Efficacy of 8 vs 4 Sessions Mindfulness-based Programs in a Non-clinical Population: a Controlled Study
Brief Title: Efficacy of 8 vs 4 Sessions Mindfulness-based Programs in a Non-clinical Population
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Javier Garcia Campayo, Dr, Hospital Miguel Servet
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: PI12/00134
Record Dates: First submitted 2015-12-18; First posted 2015-12-31 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- standard 8-weeks MBSR (Experimental): 8-week program
  Interventions: Behavioral: standard 8-weeks MBSR
- 4-week shortened MBSR (Experimental): Short 4 sessions intervention
  Interventions: Behavioral: 4-week shortened MBSR
- Control Group (No Intervention): control group: No intervention

INTERVENTIONS:
Behavioral: standard 8-weeks MBSR — A 8 weekly sessions of 120 min based on the standard protocol of Kabat Zinn was performed. The adapted program did not include a one-day retreat in silence, but one session in silence plus extra kindly awareness (compassion-based) and value-based exercises. Home practice was not systematically assessed, but recommended to be of 45min per day, most of the days. It was administered by a trained (3-y experience) and certified MBSR teacher (MMPD).
  Arms: standard 8-weeks MBSR
Behavioral: 4-week shortened MBSR — This protocol was made up of 4 sessions of 120 mn administered by the same trained MBSR programme therapist to avoid variables associated to the therapist. The rationale behind the shortened version of MBSR was to keep the core content and practices of the program, in fewer sessions: raisin exercise (experiential concept of mindfulness); and main anchors of attention (breathing, body sensations, body movements).
  Arms: 4-week shortened MBSR

SUMMARY:
The aim of this study was to assess and compare the efficacy of a standard 8-weeks protocol based on the Mindfulness Based Stress Reduction MBSR program versus a 4-week shortened version of the protocol in the improvement of wellbeing variables in a non-clinical population in Spain. The investigators initial hypothesis was that both protocols are efficacious but the standard 8-week performs better that the short one.

ELIGIBILITY:
Inclusion Criteria:

* be adult (18-y or older);
* willingness to participate in the study and signing informed consent;
* ability to understand and write Spanish.

Exclusion Criteria:

* have an acute clinical or psychiatry condition;
* have no previous experience with mindfulness or other type of contemplative or mind-boy practices such as yoga, taichi or chikung.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | baseline
Hospital Anxiety and Depression Scale (HADS) change from baseline | post-treatment 8 weeks from baseline in 8 weeks intervention group
Hospital Anxiety and Depression Scale (HADS) change from baseline | post-treatment 4 weeks from baseline in 4 weeks intervention group
Hospital Anxiety and Depression Scale (HADS) change from baseline | six-months follow-up

SECONDARY OUTCOMES:
Mindful Attention Awareness Scale (MAAS) | baseline, post-treatment 8 weeks from baseline in 8 weeks intervention group, post-treatment 4 weeks from baseline in 4 weeks intervention group, and six-months follow-up
Five Facets Mindfulness Questionnaire (FFMQ) | baseline, post-treatment 8 weeks from baseline in 8 weeks intervention group, post-treatment 4 weeks from baseline in 4 weeks intervention group, and six-months follow-up
Self-Compassion Scale (SCS) | baseline, post-treatment 8 weeks from baseline in 8 weeks intervention group, post-treatment 4 weeks from baseline in 4 weeks intervention group, and six-months follow-up
The Positive and Negative Affect Scale (PANAS) | baseline, post-treatment 8 weeks from baseline in 8 weeks intervention group, post-treatment 4 weeks from baseline in 4 weeks intervention group, and six-months follow-up
Connor-Davidson Resilience Scale (10-item CD-RISC) | baseline, post-treatment 8 weeks from baseline in 8 weeks intervention group, post-treatment 4 weeks from baseline in 4 weeks intervention group, and six-months follow-up

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Demarzo M, Montero-Marin J, Puebla-Guedea M, Navarro-Gil M, Herrera-Mercadal P, Moreno-Gonzalez S, Calvo-Carrion S, Bafaluy-Franch L, Garcia-Campayo J. Efficacy of 8- and 4-Session Mindfulness-Based Interventions in a Non-clinical Population: A Controlled Study. Front Psychol. 2017 Aug 8;8:1343. doi: 10.3389/fpsyg.2017.01343. eCollection 2017. PMID 28848465